CLINICAL TRIAL: NCT07288060
Title: The Effect of Mulligan Mobilisation and Graded Motor Imagery Therapy on Proprioception in Distal Radius Fractures
Brief Title: The Effect of Mulligan and GMI on Distal Radius Proprioception
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Collaborators: Biruni University (Other); Istanbul University (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Barış CELBEK, Lecturer, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04.04.2025/07; 424S042 (Other Grant/Funding Number: TUBİTAK)
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Distal Radial Fracture; Rehabilitation; Mulligan Mobilization; Motor Imagery Training; Physical Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional physiotherapy (Active Comparator): This group of participants will receive only standard care, defined as conventional physiotherapy, during their rehabilitation process following distal radius fracture surgery. The treatment program will commence at the 6th week post-surgery and will be applied twice a week for 6 weeks (totaling 12 sessions), with each session lasting an average of 30-35 minutes. Conventional physiotherapy includes joint range of motion exercises (flexion, extension, ulnar/radial deviation for the wrist; supination/pronation for the elbow) for 10 repetitions. Strengthening exercises, utilizing Theraband for wrist movements (10 repetitions) and Powerweb/Theraputty for grip strength (10 repetitions), will be applied, with resistance levels set at approximately 60-70% of the 1 Repetition Maximum method. Additionally, Closed Kinetic Chain exercises (wall press, plyometric wall push-ups, crawling, and push-ups after week 5) will be incorporated starting from the 3rd week of conventional treatment.
  Interventions: Other: Conventional Physiotherapy
- Mulligan Mobilisation Group (Experimental): The Mulligan Group will receive Mobilization With Movement (Mulligan MWM) techniques in addition to conventional physiotherapy, aiming to achieve pain-free movement by correcting the "positional fault" in the joint. The treatment will be administered for 6 weeks starting from the 6th week post-surgery, with 2 sessions per week (totaling 12 sessions) , and the MWM component will last approximately 15-20 minutes. MWM techniques, which must be performed pain-free, are initiated with the lateral glide of the carpal row and include continuous lateral glide to improve wrist flexion and extension. Furthermore, MWM of the distal and proximal radioulnar joint to improve supination will be added to the program starting from the 3rd week. Each mobilization is applied as 3 sets of 10 repetitions , with a rest period of 15-20 seconds between sets. To ensure continuous pain-free movement, patients will also be taught self-mobilization (10 repetitions) to be performed at home.
  Interventions: Other: Conventional Physiotherapy; Other: Mulligan Mobilisation
- Graded motor imagery(GMI) Group (Experimental): The Graded Motor Imagery (GMI) Group will implement a three-phase protocol aimed at supporting functional recovery by increasing neuroplasticity, in addition to conventional physiotherapy. The treatment will begin at the 6th week post-surgery and will be administered for 6 weeks at 2 sessions per week (12 sessions total), with the GMI component lasting approximately 15-20 minutes. The protocol is designed so that each of the three phases lasts one to two weeks due to immobilization constraints. Phase 1 (Lateralization Training) (the first 2 weeks) involves the patient correctly and quickly identifying whether presented images are of the right or left hand. Phase 2 (Explicit Motor Imagery) (the remaining 4 weeks) requires the patient to visualize movements of the affected wrist in various positions mentally, a process that is tracked via a dedicated website.Finally, during Phase 3 (Mirror Therapy), the patient moves the unaffected hand while observing its reflection, creating the illus
  Interventions: Other: Conventional Physiotherapy; Other: Graded Motor Imagery (GMI)

INTERVENTIONS:
Other: Conventional Physiotherapy — Patients receive the standard physical therapy program only.
Other: Mulligan Mobilisation — In addition to conventional therapy, Mobilization With Movement (MWM) techniques are applied, focusing on achieving pain-free motion. These techniques include lateral glides of the carpal row and wrist flexion/extension/supination movements, performed in 3 sets of 10 repetitions, and patients are taught self-mobilization.
  Arms: Mulligan Mobilisation Group
Other: Graded Motor Imagery (GMI) — This arm adds a three-phase protocol designed to target neuroplasticity. The protocol includes: Lateralization (right/left hand recognition), Explicit Motor Imagery (mental visualization of movement), and Mirror Therapy. The second phase is uniquely tracked via an internet-based platform for home exercises, which records response times and accuracy
  Arms: Graded motor imagery(GMI) Group

SUMMARY:
Distal radius fractures are common in the elderly population and clinical findings after treatment include limitation of joint motion, pain, and muscle weakness. Physical therapy modalities include exercises, physical agents, and manual therapy techniques. The Mulligan Concept-specific mobilization with movement (MWM) technique improves joint movement by reducing pain and is effective in musculoskeletal disorders. Graded motor imagery activates the motor system, increases neuroplasticity, and promotes functional recovery.

It has been observed that proprioception is impaired after distal radius fracture, affecting muscle tone and postural reflexes. Our study will examine proprioception measurements with an electrogonometer (K Force Sens) and universal goniometer and the effectiveness of MWM and progressive motor imagery treatments.

The study is designed as a one-blind randomized study and a total of 33 patients between the ages of 25-65 who were treated with volar plate screws after distal radius fracture will be included. Patients will be randomized as 11 people and one group will be treated with Mulligan Mobilisation in addition to conventional physiotherapy and the other group will be treated with Graded motor imagery techniques in addition to conventional physiotherapy. The control group will receive only conventional physiotherapy.

Clinical Follow-up Form, Proprioception, Kinesiophobia, Hand Grip strength, Muscle strength, Pain, and functional evaluations will be performed 2 times in total, just before the patient starts physical therapy after surgery and at the end of the 6-week treatment.

A goniometer and electrogoniometer will be used to measure proprioception. Visual Analogue Scale (VAS) and algometer will be used to determine the pain assessment. Jamar's hand grip strength meter and Digital Handheld Dynamometer will be used for muscle strength assessment. Tampa Kinesiophobia Scale will be used to measure the level of kinesiophobia. Patient Rated Wrist/Hand Evaluation (PRWHE) will be used to evaluate the functionality of the patients.

Proprioception evaluation in the upper extremity is limited in the literature, and it will be an original study to examine the relationship between the two measurements after distal radius fracture surgery; in addition, it will be the first study to examine graded motor imagery and mulligan Mobilisation in terms of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 65 years
* Clinical diagnosis of distal radius fracture
* Indicated for surgical treatment
* Surgical fixation performed using plate and screw technique
* Willing and able to provide informed consent and participate in the study

Exclusion Criteria:

* Inability to read or write
* Presence of additional orthopedic, neurological, or cardiovascular disorders
* History of surgery involving the ipsilateral upper extremity within the past 6 months
* Visual or hearing impairment that would interfere with adherence to treatment or study assessments

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 33 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Tampa Scale of Kinesiophobia (TSK) | From the start of physiotherapy (approximately 6 weeks post-surgery) to the end of the 6-week treatment period.
  The Tampa Scale of Kinesiophobia (TSK) is a self-report measure developed to assess the fear of pain related to movement in patients with musculoskeletal pain. It consists of 17 questions designed to measure the fear of movement and re-injury. The scale utilizes a 4-point Likert scoring system (1 = strongly disagree, 4 = strongly agree). The items are grouped into two distinct factors: activity avoidance and somatic focus. The TSK is commonly used in distal radius fracture cases to assess general fear of movement.
Proprioception Assessment (Joint Position Sense) | From the start of physiotherapy (approximately 6 weeks post-surgery) to the end of the 6-week treatment period.
  Application in Your Study: In your project, this assessment will be performed using both a universal goniometer and an electrogoniometer (K Force Sens).The patient is asked to memorize a target angle (20 extension) and then actively reproduce it, with the difference between the target angle and the measured angle recorded as the degree of error.

SECONDARY OUTCOMES:
Pain Assessment | From the start of physiotherapy (approximately 6 weeks post-surgery) to the end of the 6-week treatment period.
  Visual Analog Scale (VAS) Used to rate the severity of the patient's pain. It typically consists of a 100 mm line with two descriptors representing extreme pain intensity (e.g., no pain and worst possible pain) at either end. Patients mark their intensity on the line, and the score is measured as the distance from the "no pain" end.
Pressure Pain Threshold (PPT) | From the start of physiotherapy (approximately 6 weeks post-surgery) to the end of the 6-week treatment period.
  Algometer (Baseline dolorimeter 66 pound) Used as an objective method to measure the pressure pain threshold on the patient's wrist. Measurements are recorded in kilograms (kg). The test is 10 seconds long with gradually increasing pressure. Assessment points include the lateral epicondyle, medial epicondyle, ulnar styloid, and radial head.
Functionality & Disability | From the start of physiotherapy (approximately 6 weeks post-surgery) to the end of the 6-week treatment period.
  Patient-Rated Wrist/Hand Evaluation (PRWHE) Used to assess the patient's functionality. It is a subjective outcome measure consisting of 15 questions that determine the level of pain and disability in hand/wrist problems. It includes pain and function subscales, and sections for specific and daily activities. Total score is calculated out of 100, with a higher score indicating greater disability.
Grip Strength (Gross) | From the start of physiotherapy (approximately 6 weeks post-surgery) to the end of the 6-week treatment period.
  Jamar Hand Dynamometer considered the gold standard for measuring hand grip strength, highly reliable, and recommended by the American Society of Hand Therapists (ASHT). The measurement is taken in a standard position (seated, shoulder adducted/neutral rotation, elbow 90^\circ$ flexion, forearm mid-rotation/supported, wrist neutral). The average of 3 measurements, with 1-minute rests between each, is recorded.
Specific Muscle Strength | From the start of physiotherapy (approximately 6 weeks post-surgery) to the end of the 6-week treatment period.
  Digital Handheld Dynamometer Used to evaluate the strength of the wrist flexor, extensor, ulnar, and radial deviation muscles. The device provides objective data and records measurements in kilograms (kg) over a 10-second resistance test.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydın University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No